CLINICAL TRIAL: NCT03027024
Title: Clinical Study to Investigate Visual Performance of Hydrophobic Trifocal IOL: FineVision HP
Brief Title: Clinical Study to Investigate Visual Performance of IOL: FineVision HP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHY 1602
Record Dates: First submitted 2017-01-16; First posted 2017-01-20 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Cataract; Lens Opacity
Keywords: Intraocular Lens; trifocal; cataract; PhysIOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IOL Implantation (Experimental): Implantation of IOL: PhysIOL POD F GF
  Interventions: Device: Implantation of IOL: PhysIOL POD F GF

INTERVENTIONS:
Device: Implantation of IOL: PhysIOL POD F GF — Implantation of trifocal IOL POD F GF consisting of hydrophobic material
  Other Names: PhysIOL HP

SUMMARY:
This is a prospective, non-randomised, controlled, single-surgeon, single-center post-market clinical follow up study whereby patient undergoing routine cataract surgery will have bilateral implantation of a recently introduced TGA (Therapeutics Goods Authority, Australia) approved trifocal intraocular lens FineVision Evo (PhysIOL, Liège, Belgium). The primary and secondary effectiveness data for visual acuity, defocus curves, contrast sensitivity and any adverse events will be collected.

DETAILED DESCRIPTION:
Subjects participating in the trial will attend a total of 8 study visits (1 preoperative, 2 operative and 5 postoperative) over a period of 3 months, same as the surgeon's standard follow up protocol for bilateral cataract surgery with IOL implantation. Subjects would have the option for unscheduled visits if required medically.

Primary endpoint data will be collected at the final visit. Data analyses will be done in the end to support the study publication plan.

ELIGIBILITY:
Inclusion Criteria:

* Cataracteous eyes with no comorbidity
* Spontaneously emitting the desire for spectacle independence after surgery and with realistic expectation.
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Signed informed consent

Exclusion Criteria:

* Unrealistic expectation
* Irregular astigmatism
* Regular corneal astigmatism >0.75 D on one or both eyes as measured by an automatic keratometer (regularity determined by the topography of the keratometry)
* Difficulty for cooperation (distance from their home, general health condition)
* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus (with retinopathy), immunocompromised, glaucoma etc…)
* Any ocular comorbidity
* History of ocular trauma or prior ocular surgery including refractive procedures
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, chronic Uveitis, Marfan's syndrome)
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic/scotopic conditions)
* Complicated surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
binocular Distance Corrected Near Visual Acuity (DCNVA) | 3 months postoperative
  measured in logMAR

SECONDARY OUTCOMES:
monocular and binocular Uncorrected Distance Visual Acuity (UDVA) | 3 months postoperative
  measured in logMAR
monocular and binocular Corrected Distance Visual Acuity (CDVA) | 3 months postoperative
  measured in logMAR
monocular and binocular Uncorrected Intermediate Visual Acuity (UIVA) | 3 months postoperative
  measured in logMAR
monocular and binocular Distance Corrected Intermediate Visual Acuity (DCIVA) | 3 months postoperative
  measured in logMAR
monocular and binocular Uncorrected Near Visual Acuity (UNVA) | 3 months postoperative
  measured in logMAR
monocular and binocular Distance Corrected Near Visual Acuity (DCNVA) | 3 months postoperative
  measured in logMAR
Contrast Sensitivity (mesopic and photopic) | 3 months postoperative
  measured in logCS

CONTACTS AND LOCATIONS:
Overall Officials: Uday Bhatt, MD, Principal Investigator — Vision Eye Institute - Footscray
Locations (1):
- Vision Eye Institute, Footscray, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No